CLINICAL TRIAL: NCT04433715
Title: Identification of the Urogenital Distress Inventory-6 and the Incontinence Impact Questionnaire-7 Cutoff Scores in Urinary Incontinent Women
Brief Title: Identification of the UDI-6 and the IIQ-7 Cutoff Scores in Urinary Incontinent Women
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Katarzyna Skorupska, Principal Investigator, Medical University of Lublin
Other Study IDs: 01/2020
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Quality of Life; Urinary Incontinence,Stress; Urinary Incontinence
Keywords: Incontinence Impact Questionnaire-7; Urogenital Distress Inventory-6
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with UI symptoms: All participants completed all three questionnaires: ICIQ-SF, UDI-6 and IIQ-7.
  Interventions: Diagnostic Test: ICIQ-SF; Diagnostic Test: UDI-6; Diagnostic Test: IIQ-7
- patients without UI symptoms: All participants completed all three questionnaires: ICIQ-SF, UDI-6 and IIQ-7.
  Interventions: Diagnostic Test: ICIQ-SF; Diagnostic Test: UDI-6; Diagnostic Test: IIQ-7

INTERVENTIONS:
Diagnostic Test: ICIQ-SF — All participants completed ICIQ-SF,
Diagnostic Test: UDI-6 — All participants completed UDI-6
Diagnostic Test: IIQ-7 — All participants completed IIQ-7

SUMMARY:
Purpose Urogenital Distress Inventory-6 (UDI-6), Incontinence Impact Questionnaire-7 (IIQ-7) and The International Consultation on Incontinence (ICIQ-SF) Short Form are used to diagnose individuals with urinary incontinence (UI) and to assess the impact of the dysfunction on patient quality of life. While ICIQ-SF has fixed cutoff values - UDI-6 and IIQ-7 do not. We aimed to find the cutoff scores for UDI-6 and IIQ-7 in women with UI.

Methods The study involved 205 women aged between 31 and 83 years - 155 with, and 50 without UI symptoms. All participants completed all three questionnaires: ICIQ-SF, UDI-6 and IIQ-7. Patients were categorized according to their ICIQ-SF scores, as symptomatic ICIQ-SF ≥6 (n=134) and asymptomatic ICIQ < 6 (n=60). The Receiver Operating Characteristics (ROC) curve was used to test how well UDI-6 allowed a discrimination between patients suffering from UI and those who do not. AUC (Area under Curve) statistic was calculated to measure the UDI-6 and IIQ-7 Total Score efficiency.

DETAILED DESCRIPTION:
Purpose Urogenital Distress Inventory-6 (UDI-6), Incontinence Impact Questionnaire-7 (IIQ-7) and The International Consultation on Incontinence (ICIQ-SF) Short Form are used to diagnose individuals with urinary incontinence (UI) and to assess the impact of the dysfunction on patient quality of life. While ICIQ-SF has fixed cutoff values - UDI-6 and IIQ-7 do not. We aimed to find the cutoff scores for UDI-6 and IIQ-7 in women with UI.

Methods The study involved 205 women aged between 31 and 83 years - 155 with, and 50 without UI symptoms. All participants completed all three questionnaires: ICIQ-SF, UDI-6 and IIQ-7. Patients were categorized according to their ICIQ-SF scores, as symptomatic ICIQ-SF ≥6 (n=134) and asymptomatic ICIQ < 6 (n=60). The Receiver Operating Characteristics (ROC) curve was used to test how well UDI-6 allowed a discrimination between patients suffering from UI and those who do not. AUC (Area under Curve) statistic was calculated to measure the UDI-6 and IIQ-7 Total Score efficiency.

ELIGIBILITY:
Inclusion Criteria:

* UI symptoms

Exclusion Criteria:

* lack of consent, oncological diseases

Ages: 31 Years to 83 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study involved a total of 205 women aged between 31 and 83 years who were recruited from women attending the Gynecological Outpatient Clinic due to UI symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
patients with sympthomatic UI- ICIQ-SF ≥6 | 01.03.2016-30.06.2016
  symptomatic ICIQ-SF ≥6
asymphomatic patients ICIQ-SF<6 | 01.03.2016-30.06.2016
  ICIQ<6

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Rechberger, Study Director — Medical University of Lublin
Locations (1):
- Katarzyna Skorupska, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Yes
We would like to share UDI-6 and IIQ-7 cutoff scores
Supporting Information: Study Protocol
Time Frame: 2020
Access Criteria: email co PI kasiaperzylo@hotmail.com

REFERENCES:
- [Derived] Skorupska K, Grzybowska ME, Kubik-Komar A, Rechberger T, Miotla P. Identification of the Urogenital Distress Inventory-6 and the Incontinence Impact Questionnaire-7 cutoff scores in urinary incontinent women. Health Qual Life Outcomes. 2021 Mar 16;19(1):87. doi: 10.1186/s12955-021-01721-z. PMID 33726776